CLINICAL TRIAL: NCT01754727
Title: Impact of Adalimumab (Humira®) Therapy on Selected Health Care Resource Utilization and Sick Leave in Patients With Ankylosing Spondylitis in Clinical Practice
Acronym: IDEA
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-682
Record Dates: First submitted 2012-12-19; First posted 2012-12-21 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Effectiveness; Post-marketing observational study (PMOS); Adalimumab; Humira®
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Ankylosing Spondylitis (AS): Participants with ankylosing spondylitis treated with adalimumab in routine clinical practice.

SUMMARY:
The purpose of this study was to assess the proportion of AS patients achieving treatment response to adalimumab therapy.

DETAILED DESCRIPTION:
This post-marketing observational study (PMOS) was performed in a multi-country, multi-center, single-arm format. Data were collected prospectively and retrospectively. Adult patients with diagnosis of AS who were assigned for treatment with adalimumab (Humira®) were eligible for participation. Each patient included in this study was to be observed during his/her adalimumab treatment for a maximum of 12 month period. During this period four follow-up visits were planned for observation of the patient and documentation of data. Ideally, these visits should have been performed approximately 3 (V1), 6 (V2), 9 (V3) and 12 (V4) months after the baseline visit (V0).

ELIGIBILITY:
Inclusion Criteria:

* Had ankylosing spondylitis (AS) and was eligible to start and/or continue adalimumab therapy according to the local product label and prescription guidelines,
* Had been started on adalimumab therapy no more than one (1) month prior to the study enrollment
* Had negative result of tuberculosis (TB) screening test or was receiving tuberculosis prophylaxis as per local guidelines
* Provided written Authorization to the investigator to use and/or disclose personal and/or health data, or Informed Consent if requested by the Local Regulations

Exclusion Criteria:

- Had contraindications for the treatment with adalimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consisted of participants with ankylosing spondylitis (AS) who were treated with adalimumab as per locally approved label and prescription guidelines. The decision to be treated with adalimumab had to be independent from study inclusion.
Sampling Method: Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Iosub, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 452 participants were enrolled: 450 were in the main analysis set (MAS) population; 2 were excluded from MAS, as adalimumab treatment was not documented within this study.
Groups:
- Participants With Ankylosing Spondylitis: Participants with ankylosing spondylitis treated with adalimumab in routine clinical practice.
Period: Overall Study
Arm/Group | Participants With Ankylosing Spondylitis
Started | 452
Completed | 450
Not Completed | 2
Not completed — Adalimumab Treatment was not Documented | 2

BASELINE CHARACTERISTICS:
Population: Baseline analyses accounts for main analysis set (MAS) population (all participants who received at least 1 dose of study drug).
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 450
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age (continuous) measure analysis accounts for main analysis set (MAS) population (all participants who received at least 1 dose of study drug) with evaluable data.
  years
    number analyzed (Participants) | 447
    (all) | 42.9 (12.1)
Gender [Count of Participants; unit: Participants]
  Female | 141
  Male | 309

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 at Month 12
Description: The BASDAI score was determined using a simple, self-reported questionnaire that consists of 6 questions on disease activity. Each question is scored from 0 to 10 (0 = no symptoms, 10 = very severe symptoms). The BASDAI 50 score captures patients with 50% reduction in the BASDAI score compared to baseline as observed.
Time Frame: Month 0 (baseline) and Month 12
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 351
percentage of participants | 78.9

2. Secondary Outcome: Percentage of Participants Achieving BASDAI 50
Description: The BASDAI score was determined using a simple, self-reported questionnaire that consists of 6 questions on disease activity. Each question is scored from 0 to 10 (0 = no symptoms, 10 = very severe symptoms). The BASDAI 50 score captures patients with 50% reduction in the BASDAI score compared to baseline.
Time Frame: Month 3, Month 6 and Month 9
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 425
percentage of participants
  Month 3 (N=425) | 52.5
  Month 6 (N=395) | 68.1
  Month 9 (N=367) | 76.0

3. Secondary Outcome: Percentage of Participants Achieving At Least 2.0 Score Decrease in Ankylosing Spondylitis Disease Activity (ASDAS) Score From Baseline
Description: The ASDAS tool is a self-administered questionnaire plus an objective laboratory evaluation. The questionnaire covers disease activity, back pain, and peripheral pain/swelling assessed on a visual analogue scale (from 0 (normal) to 10 (extreme pain or disability) cm) and duration of morning stiffness on a numerical rating scale (from 0 to 10, with 0 being none and 10 representing a duration of 2 hours or longer). The laboratory parameter is a measurement of C-reactive protein (mg/L) (CRP) or erythrocyte sedimentation rate (mm/h) (ESR). Data from five variables (disease activity, back pain, duration of morning stiffness, peripheral pain/swelling, and either CRP or ESR values) are combined to yield a score ranging from 0 to no defined upper limit. Higher scores indicate higher disease activity. Clinically important improvement is defined as a change >= 1.1 units, and major improvement is defined as a change >= 2.0 units.
Time Frame: Month 3, Month 6, Month 9 and Month 12
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 424
percentage of participants
  Month 3 (N=424) | 44.3
  Month 6 (N=393) | 54.5
  Month 9 (N=364) | 63.5
  Month 12 (N=349) | 64.8

4. Secondary Outcome: Mean Change in the Number of Hospital Inpatient Days
Description: Difference in the number of hospital inpatient days during 12 months of adalimumab therapy and 12 months preceding the introduction of adalimumab therapy.
Time Frame: 12 months prior to month 0 (baseline) and 12 months prior to month 12
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 365
Days | -19.6 (45.0)

5. Secondary Outcome: Mean Change in the Number of Hospitalizations
Description: Difference in the number of hospitalizations during 12 months of adalimumab therapy and 12 months preceding the introduction of adalimumab therapy.
Time Frame: 12 months prior to month 0 (baseline) and 12 months prior to month 12
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: Number of admissions to hospital
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 376
Number of admissions to hospital | -1.9 (4.4)

6. Secondary Outcome: Mean Change in the Number of Sick Leave Days
Description: Difference in the number of sick leave days during 12 months of adalimumab therapy and 12 months preceding the introduction of adalimumab therapy (in employed subjects only)
Time Frame: 12 months prior to month 0 (baseline) and 12 months prior to month 12
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 235
Days | -27.3 (66.3)

7. Secondary Outcome: Mean Change in the Number of Sick Leaves
Description: Difference in the number of sick leaves during 12 months of adalimumab therapy and 12 months preceding the introduction of adalimumab therapy (in employed subjects only).
Time Frame: 12 months prior to month 0 (baseline) and 12 months prior to month 12
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: Number of sick leaves
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 237
Number of sick leaves | -2.1 (5.3)

8. Secondary Outcome: Mean Change in the Number of Outpatient Visits to Each Kind of Health Care Provider
Description: Difference in the number of outpatient visits to each kind of health care provider which includes general practitioner, rheumatologist, other specialists (ophthalmologist, gastroenterologist, dermatologist, physiatrist), physiotherapist and rheumatology nurse, during 12 months of adalimumab therapy and 12 months preceding the introduction of adalimumab therapy.
Time Frame: 12 months prior to month 0 (baseline) and 12 months prior to month 12
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 403
Number of visits
  Overall (N=403) | -12.1 (23.1)
  General practitioner (N=354) | -4.3 (8.7)
  Rheumatologists (N=399) | -4.4 (8.3)
  Ophthalmologist (N=313) | -1.1 (4.3)
  Gastroenterologist (N=309) | -0.6 (3.1)
  Dermatologist (N=311) | -0.4 (2.5)
  Physiatrist (N=310) | -0.5 (1.9)
  Physiotherapist (N=315) | -1.9 (10.6)
  Rheumatology nurse (N=315) | -0.5 (7.5)

9. Secondary Outcome: Mean Change From Baseline in BASDAI Score
Description: The BASDAI score was determined using a simple, self-reported questionnaire that consists of 6 questions on disease activity. Each question is scored from 0 to 10 (0 = no symptoms, 10 = very severe symptoms).
Time Frame: Month 3, Month 6, Month 9, Month 12 and Month 12 Last Observation Carried Forward (LOCF)
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 429
units on a scale
  Month 3 (N=425) | -3.1 (2.3)
  Month 6 (N=395) | -3.8 (2.4)
  Month 9 (N=367) | -4.3 (2.3)
  Month 12 (N=351) | -4.4 (2.4)
  Month 12 LOCF (N=429) | -4.0 (2.6)

10. Secondary Outcome: Mean Change From Baseline in Ankylosing Spondylitis Disease Activity (ASDAS) Score
Description: The ASDAS tool is a self-administered questionnaire plus an objective laboratory evaluation. The questionnaire covers disease activity, back pain, and peripheral pain/swelling assessed on a visual analogue scale (from 0 (normal) to 10 (extreme pain or disability) cm) and duration of morning stiffness on a numerical rating scale (from 0 to 10, with 0 being none and 10 representing a duration of 2 hours or longer). The laboratory parameter is a measurement of C-reactive protein (mg/L) (CRP) or erythrocyte sedimentation rate (mm/h) (ESR). Data from five variables (disease activity, back pain, duration of morning stiffness, peripheral pain/swelling, and either CRP or ESR values) are combined to yield a score ranging from 0 to no defined upper limit. Higher scores indicate higher disease activity. Remission is defined as ASDAS score <1.3. Clinically important improvement is defined as a change >= 1.1 units, and major improvement is defined as a change >= 2.0 units.
Time Frame: Month 3, Month 6, Month 9 and Month 12
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 428
units on a scale
  Month 3 (N=424) | -1.8 (1.3)
  Month 6 (N=393) | -2.1 (1.3)
  Month 9 (N=364) | -2.3 (1.2)
  Month 12 (N=349) | -2.4 (1.3)
  Month 12 LOCF (N=428) | -2.2 (1.4)

11. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Score
Description: The BASFI is a numeric rating scale that uses self-reported patient evaluations to measure physical function impairment caused by AS. It is a ten questions, each question was scored on a numerical rating scale that ranged from 0 (no functional impairment) to 10 (maximal impairment). The mean of the ten questions was the total BASFI score. A higher score indicates more severe impairment of functioning.
Time Frame: Month 3, Month 6, Month 9 and Month 12
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 422
units on a scale
  Month 3 (N=414) | -2.7 (2.4)
  Month 6 (N=381) | -3.5 (2.4)
  Month 9 (N=356) | -3.8 (2.3)
  Month 12 (N=339) | -4.0 (2.5)
  Month 12 LOCF (N=422) | -3.6 (2.6)

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time the participant's informed consent was received until 30 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment i.e., up to 12 months.
Description: Non serious adverse events were not collected for this study.
Arm/Group | Participants With Ankylosing Spondylitis
Serious Adverse Events (participants affected / at risk) | 19/450
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Ankylosing Spondylitis (N=450)
ANAEMIA (Blood and lymphatic system disorders) | 1
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 1
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1
ADMINISTRATION SITE RASH (General disorders) | 1
DRUG INEFFECTIVE (General disorders) | 2
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1
CYSTITIS (Infections and infestations) | 1
GINGIVITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 1
TUBERCULOSIS (Infections and infestations) | 1
TUBERCULOUS PLEURISY (Infections and infestations) | 1
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
HYPERTONIA (Nervous system disorders) | 1
ANXIETY (Psychiatric disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1
RENAL COLIC (Renal and urinary disorders) | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 2
RASH (Skin and subcutaneous tissue disorders) | 1
HYPERTENSION (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.